CLINICAL TRIAL: NCT00069836
Title: A 24 Week, Randomised, Double Blind, Parallel Study to Compare the Change in HbA1c With AVANDAMET® (8.0mg / 2.0g) Plus Insulin to Placebo Plus Insulin, in Subjects With Type 2 Diabetes Starting Insulin Therapy
Brief Title: Study Of AVANDAMET® With Or Without Insulin In Type II Diabetes Mellitus Patients. AVANDAMET® is a Registered Trademark of the GSK Group of Companies.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 712753/009
Record Dates: First submitted 2003-10-01; First posted 2003-10-03 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: AVANDAMET insulin type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rosiglitazone-metformin combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Rosiglitazone/metformin

INTERVENTIONS:
Drug: Rosiglitazone/metformin

SUMMARY:
This study was designed to test the safety and efficacy (how well it works) of AVANDAMET in combination with insulin in improving the control of blood sugar when compared with taking insulin on its own. AVANDAMET capsules contain a fixed dose of AVANDIA and metformin. Both AVANDIA and metformin are medicines which are individually licensed for the treatment of type II diabetes mellitus. Because they act in different ways, it is thought that combining them may give an increased benefit of treating diabetes and reducing blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been diagnosed with type II diabetes mellitus and not have adequate glycaemic controlled while receiving at least 1.5g of metformin.
* Patients must have a body mass index of greater than 25 kg/m2 and must not suffer from ankle swelling.

Exclusion Criteria:

* Patients cannot have any form of congestive heart failure or severe or unstable angina.
* Patients cannot be currently receiving insulin, but be prepared to begin insulin treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2003-10; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | 24 weeks

SECONDARY OUTCOMES:
Insulin dose, FPG,glycaemic responders, beta-cell function, hypoglycaemia, treatment satisfaction | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (79):
- GSK Investigational Site, Vienna, Austria
- France (19):
  - GSK Investigational Site, Roubaix, Hauts-de-France
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Bondy
  - GSK Investigational Site, Cholet
  - GSK Investigational Site, Corbeil-Essonnes
  - GSK Investigational Site, Douai
  - GSK Investigational Site, Épinay-sur-Orge
  - GSK Investigational Site, La Rochelle
  - GSK Investigational Site, Lorient
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Montbrison
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, St-Malo
  - GSK Investigational Site, Toul
  - GSK Investigational Site, Vénissieux
- Germany (40):
  - GSK Investigational Site, Hermaringen, Baden-Wurttemberg
  - GSK Investigational Site, Kippenheim, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Sinsheim, Baden-Wurttemberg
  - GSK Investigational Site, Stockach, Baden-Wurttemberg
  - GSK Investigational Site, Ilvesheim, Bavaria
  - GSK Investigational Site, Künzing, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Wallerfing, Bavaria
  - GSK Investigational Site, Falkensee, Brandenburg
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Schwedt, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Bad Kreuznach, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Schlüchtern, Hesse
  - GSK Investigational Site, Vellmar, Hesse
  - GSK Investigational Site, Hildesheim, Lower Saxony
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Bad Oeynhausen, North Rhine-Westphalia
  - GSK Investigational Site, Beckum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Viersen, North Rhine-Westphalia
  - GSK Investigational Site, Altenkirchen, Rhineland-Palatinate
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Simmern, Rhineland-Palatinate
  - GSK Investigational Site, Speyer, Rhineland-Palatinate
  - GSK Investigational Site, Saarlouis, Saarland
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freital, Saxony
  - GSK Investigational Site, Pirna, Saxony
  - GSK Investigational Site, Halberstadt, Saxony-Anhalt
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Gotha, Thuringia
  - GSK Investigational Site, Schleiz, Thuringia
- Italy (6):
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Pordenone, Friuli Venezia Giulia
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Perugia, Umbria
  - GSK Investigational Site, Padua, Veneto
  - GSK Investigational Site, Treviso, Veneto
- Spain (13):
  - GSK Investigational Site, Alcobendas/Madrid
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Cadiz
  - GSK Investigational Site, Galdakano
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Móstoles/Madrid
  - GSK Investigational Site, Pontevedra
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, Sant Joan d'Alacant
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo/Pontevedra

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Home PD, Bailey CJ, Donaldson J, Chen H, Stewart MW. A double-blind randomized study comparing the effects of continuing or not continuing rosiglitazone + metformin therapy when starting insulin therapy in people with Type 2 diabetes. Diabet Med. 2007 Jun;24(6):618-25. doi: 10.1111/j.1464-5491.2007.02141.x. Epub 2007 Apr 2. PMID 17403121
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 712753/009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 712753/009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 712753/009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 712753/009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 712753/009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 712753/009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 712753/009 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register